CLINICAL TRIAL: NCT00530530
Title: ASP8825 Phase ⅡStudy-A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of ASP8825 in Patients With Restless Legs Syndrome
Brief Title: ASP8825 - Study in Patients With Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8825-CL-0003
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Restless Legs Syndrome
Keywords: ASP8825; Restless legs Syndrome; XP13512
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Dose 1
  Interventions: Drug: ASP8825
- 2 (Experimental): Dose 2
  Interventions: Drug: ASP8825
- 3 (Experimental): Dose 3
  Interventions: Drug: ASP8825
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8825 — oral
  Other Names: XP13512
  Arms: 1; 2; 3
Drug: Placebo — oral
  Arms: 4

SUMMARY:
To demonstrate the superiority of ASP8825 over placebo and the dose response in patients with restless legs syndrome

DETAILED DESCRIPTION:
Three doses of ASP8825 are compared to placebo in efficacy and safety point of view in patients with restless legs syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients with RLS, based on the International RSL Study Group Diagnostic Criteria
* History of RLS symptoms at least 15 nights in the prior month or, if on treatment, this frequency of symptoms before treatment was started
* Documented RLS symptoms for at least 4 of the 7 consecutive evenings/ nights during the baseline study period

Exclusion Criteria:

* A sleep disorder (e.g., sleep apnea) that may significantly affect the assessment of RLS
* A history of RLS symptom augmentation or end-of-dose rebound with previous dopamine agonist treatment
* Neurologic disease or movement disorder (e.g., diabetic neuropathy, Parkinson's Disease, Multiple Sclerosis, dyskinesias and dystonias

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The change of the International Restless Legs Syndrome rating scale score | 12 weeks

SECONDARY OUTCOMES:
Investigator-related Clinical Global Impression of Improvement | 12 weeks
Patient- related Clinical Global Impression of Improvement | 12 weeks
The Pittsburgh sleep quality index | 12 weeks
The SF-36 Health Survey | 12 weeks
The Restless Legs Syndrome QOL Questionnaire | 12 weeks
The Medical Outcomes Study sleep scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chugoku
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Tōhoku

REFERENCES:
- [Derived] Inoue Y, Hirata K, Uchimura N, Kuroda K, Hattori N, Takeuchi M. Gabapentin enacarbil in Japanese patients with restless legs syndrome: a 12-week, randomized, double-blind, placebo-controlled, parallel-group study. Curr Med Res Opin. 2013 Jan;29(1):13-21. doi: 10.1185/03007995.2012.746217. Epub 2012 Nov 30. PMID 23121149